CLINICAL TRIAL: NCT03744897
Title: Effect of Hypnosis Combined to Transcranial Direct Stimulation in Cortical Activity and Pain Perception in Healthy Females
Brief Title: Effect of Hypnosis Combined to Transcranial Direct Stimulation in Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Principal Investigator, Wolnei Caumo, Professor of Surgery Department - School of Medicine - Head of HCPA Pain and Palliative Care Outpatient, Hospital de Clinicas de Porto Alegre
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 16-0635
Record Dates: First submitted 2017-09-21; First posted 2018-11-19 (Actual); Last update posted 2018-11-26 (Actual); Status verified 2018-11

CONDITIONS: Pain Perception; Pain Acute
Keywords: pain perception; tDCS; Hypnosis; cortical activity
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Intervention Model Description: 1. Hypnotic analgesia + a-tDCS
  2. Hypnotic analgesia + s-tDCS
  3. Hypnotic analgesia
  4. a-tDCS
Who Masked: Participant, Outcomes Assessor
Masking Description: Subjects are blinded to wether group they will be allocated Assessor will be blinded and the investigator not involved in subjects assessment will perform the hypnosis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Hypnotic analgesia (Experimental): Intervention:
  - Subjects will receive hypnotic analgesia
  Interventions: Behavioral: Hypnotic analgesia
- a-tDCS (Experimental): Intervention: transcranial direct current stimulation - tDCS
  * active tDCS stimulation
  * montage: bilateral DLPFC anodal/left and cathodal/right
  * current:2 milliamps
  * time: 20 minutes
  Interventions: Behavioral: Hypnotic analgesia; Device: s-tDCS
- s-tDCS (Sham Comparator): Sham comparator: transcranial direct current stimulation - tDCS
  * sham tDCS stimulation
  * montage: bilateral DLPFC anodal/left and cathodal/right
  * current: 0 milliamps
  * time: 20 minutes
  Interventions: Device: a-tDCS; Other: Hypnotic analgesia + a-tDCS
- Hypnotic analgesia + a-tDCS (Experimental): Intervention:
  * hypnotic analgesia
  * active tDCS stimulation
  * montage: bilateral DLPFC anodal/left and cathodal/right
  * current:2 milliamps
  * time: 20 minutes
  Interventions: Other: Hypnotic analgesia + a-tDCS

INTERVENTIONS:
Behavioral: Hypnotic analgesia — Subjects will receive hypnotic analgesia during 20 minutes
  Arms: Hypnotic analgesia; a-tDCS
Device: a-tDCS — Subjects will receive transcranial direct stimulation over bilateral DLPFC left/anode right/cathodal, 2mA, 20 minutes
  Arms: s-tDCS
Other: Hypnotic analgesia + a-tDCS — Subjects will receive hypnotic analgesia associated to transcranial direct stimulation over bilateral DLPFC left/anode right/cathodal, 2mA, 20 minutes
  Arms: Hypnotic analgesia + a-tDCS; s-tDCS
Device: s-tDCS — Subjects will receive sham transcranial direct stimulation over bilateral DLPFC left/anode right/cathodal, 0mA, 20 minutes
  Arms: a-tDCS

SUMMARY:
Pain is a public health condition, which causes great functional disability. Its consequences pervade the personal and social life of the patient, leading to significant changes in their interpersonal relationships, including work, family and social spheres, reducing the ability to perform daily activities. Conventional treatment modalities have been show a very poor therapeutic response, in that most individuals end up becoming polymedicated patients and refractory to treatment. Among non-pharmacological techniques with promising analgesic effects it includes both the hypnotic analgesia and the transcranial stimulation of direct current (tDCS).

DETAILED DESCRIPTION:
Introduction: Pain is a public health condition, which causes great functional disability. Its consequences pervade the personal and social life of the patient, leading to significant changes in their interpersonal relationships, including work, family and social spheres, reducing the ability to perform daily activities. Conventional treatment modalities have been show a very poor therapeutic response, in that most individuals end up becoming polymedicated patients and refractory to treatment. Among non-pharmacological techniques with promising analgesic effects it includes both the hypnotic analgesia and the transcranial stimulation of direct current (tDCS). Objective: To evaluate the synergistic effect of hypnotic analgesia associated with tDCS under metabolites parameters and pain levels in healthy individuals before a nociceptive stimulation pattern. Methods: it will be performed a blinded crossover sham controlled randomized clinical trial. It will be included 32 woman healthy subjects, Susceptible to the hypnosis technique according to the Scale of Hypnotic Susceptibility (WSGC) Scale of Hypnotic Scale score. aged 18 to 65. They will be allocated in one of the following groups: active tDCS + hypnotic analgesia, sham tDCS + hypnotic analgesia, hypnotic analgesia and tDCS . After a 7 days interval, the groups will be crossed in order to receive the opposite intervention of the first week. The primary endpoints will be the electrophysiological brain parameters, such as changes in the Theta, Alpha and Gamma waves, as measured by EEG. The secondary endpoints will be the level of pain, measured against nociceptive induced by the cold test and stimuli standardized pressure through algometry pressure and power down system modulatory pain, pain using the subject test - CPM - task. The intra and inter-group comparisons will be made by means of two-way ANOVA followed by Bonferroni. A p significance level of <0.05 was established. Expected results: This study hypothesizes that a synergistic effect of analgesic techniques in pain levels in healthy subjects compared to isolated character.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Female
* 11 years of schooling
* 12 cut-off at Waterloo-Stanford Group C (WSGC)

Exclusion Criteria:

* hearing loss subjects
* formal contraindication to tDCS (pregnancy, deep brain device, epilepsy, seizure)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2017-07-18 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Change in Alpha waves | 60 minutes
  Variations in the alpha waves power from post to pre-intervention using electroencephalography during a cold pressor test
Change in Theta waves | 60 minutes
  Variations in the theta waves power from post to pre-intervention using electroencephalography during a cold pressor test

SECONDARY OUTCOMES:
Change in beta waves | 60 minutes
  Variations in the beta waves power from post to pre-intervention using electroencephalography during a cold pressor test
Change in gamma waves | 60 minutes
  Variations in the gamma waves power from post to pre-intervention using electroencephalography during a cold pressor test
Change in delta waves | 60 minutes
  Variations in the delta waves power from post to pre-intervention using electroencephalography during a cold pressor test
Change in Heat thermal threshold | 60 minutes
  The measure will be assessed by Quantitative Sensorial Test - QST, in which a thermode delivers a heat stimulus of increasing magnitude. Heat thermal threshold (HTT) is the averaged temperature for 3 stimuli where participant indicates the first heat sensation.
Change in Heat pain threshold | 60 minutes
  The measure will be assessed by Quantitative Sensorial Test - QST, in which a thermode delivers a heat stimulus of increasing magnitude. Heat pain threshold (HPT) is the averaged temperature for 3 stimuli where participant indicates the first heat pain sensation.
Change in Heat pain tolerance | 60 minutes
  The measure will be assessed by Quantitative Sensorial Test - QST, in which a thermode delivers a heat stimulus of increasing magnitude. Heat pain tolerance (HPTo) is the temperature for the stimulus where participant indicates the maximum pain tolerance.
Change in Numeric pain scale during CPM task | 60 minutes
  The measure will be assessed by the conditioned pain modulation (CPM) task in which an ice cold water (0 a 1 degrees Celsius) is the conditioning stimulus presented to the left hand and a moderate heat pain stimulus from the QST to the contralateral hand. The measure consists of the response using a numeric pain scale (0 - 10) for the heat pain stimulus during the CPM task.
Change in Cold Pressor Test 0 to 1 degree Celsius - time | 60 minutes
  Participant puts his right hand in an ice cold water (0 a 1 degrees Celsius). Measure consists of the time (in seconds) the participant keeps his hand in the water the maximum he could tolerance.
Change in Cold Pressor Test 10 degree Celsius - time | 60 minutes
  Participant puts his right hand in an ice cold water (10 degrees Celsius). Measure consists of the time (in seconds) the participant keeps his hand in the water the maximum he could tolerate.
Change in Cold Pressor Test 10 degree Celsius - pain | 60 minutes
  Participant puts his right hand in an ice cold water (10 degrees Celsius). Measure consists of the response to a numeric pain scale (0 to 10) to the pain sensation when the participant withdraw his hand from the water.

CONTACTS AND LOCATIONS:
Overall Officials: Wolnei Caumo, MD. PhD, Principal Investigator — Federal University of Rio Grande do Sul
Locations (2):
- Brazil (2):
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital de Clinicas e Porto Alegre (HCPA), Porto Alegre, Rio Grande do Sul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jensen MP, Sherlin LH, Fregni F, Gianas A, Howe JD, Hakimian S. Baseline brain activity predicts response to neuromodulatory pain treatment. Pain Med. 2014 Dec;15(12):2055-63. doi: 10.1111/pme.12546. Epub 2014 Oct 7. PMID 25287554
- [Result] Jensen MP, Day MA, Miro J. Neuromodulatory treatments for chronic pain: efficacy and mechanisms. Nat Rev Neurol. 2014 Mar;10(3):167-78. doi: 10.1038/nrneurol.2014.12. Epub 2014 Feb 18. PMID 24535464
- [Result] Vanegas H, Schaible HG. Descending control of persistent pain: inhibitory or facilitatory? Brain Res Brain Res Rev. 2004 Nov;46(3):295-309. doi: 10.1016/j.brainresrev.2004.07.004. PMID 15571771
- [Result] Foerster AS, Rezaee Z, Paulus W, Nitsche MA, Dutta A. Effects of Cathode Location and the Size of Anode on Anodal Transcranial Direct Current Stimulation Over the Leg Motor Area in Healthy Humans. Front Neurosci. 2018 Jul 4;12:443. doi: 10.3389/fnins.2018.00443. eCollection 2018. PMID 30022928
- [Result] Fregni F, Boggio PS, Mansur CG, Wagner T, Ferreira MJ, Lima MC, Rigonatti SP, Marcolin MA, Freedman SD, Nitsche MA, Pascual-Leone A. Transcranial direct current stimulation of the unaffected hemisphere in stroke patients. Neuroreport. 2005 Sep 28;16(14):1551-5. doi: 10.1097/01.wnr.0000177010.44602.5e. PMID 16148743
- [Derived] Beltran Serrano G, Pooch Rodrigues L, Schein B, Zortea M, Torres ILS, Fregni F, Caumo W. The Hypnotic Analgesia Suggestion Mitigated the Effect of the Transcranial Direct Current Stimulation on the Descending Pain Modulatory System: A Proof of Concept Study. J Pain Res. 2020 Sep 16;13:2297-2311. doi: 10.2147/JPR.S253747. eCollection 2020. PMID 32982393
- [Derived] Beltran Serrano G, Rodrigues LP, Schein B, Souza A, Torres ILS, da Conceicao Antunes L, Fregni F, Caumo W. Comparison of Hypnotic Suggestion and Transcranial Direct-Current Stimulation Effects on Pain Perception and the Descending Pain Modulating System: A Crossover Randomized Clinical Trial. Front Neurosci. 2019 Jun 26;13:662. doi: 10.3389/fnins.2019.00662. eCollection 2019. PMID 31297046